CLINICAL TRIAL: NCT06960499
Title: Predictors of Physical Activity in Adult Patients With Hemophilic Arthropathy. A Multicenter Cross-sectional Cohort Study
Brief Title: Predictors of Physical Activity in Adult Patients With Hemophilic Arthropathy
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, Universidad Católica San Antonio de Murcia
Other Study IDs: HeActivity
Record Dates: First submitted 2025-04-28; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Hemophilia
Keywords: Hemophilia; Physical activity; Kinesiophobia; Functionality; Joint pain
MeSH Terms: conditions — Hemophilia A; Motor Activity; Kinesiophobia; Arthralgia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observacional group: Patients with hemophilia A or B, of legal age, with a medical diagnosis of severe phenotype of the disease and hemophilic arthropathy in the lower limbs.
  Interventions: Other: Surveys

INTERVENTIONS:
Other: Surveys — No intervention will be carried out in this study; the recruited patients will only complete the questionnaires provided below

SUMMARY:
Introduction. The development of hemophilic arthropathy causes degenerative joint damage that leads to functional impairment, limiting physical activity and causing disability in patients with hemophilia.

Objectives. i) To assess the level of physical activity in patients with hemophilia; ii) To identify the best predictive model for physical activity in adult patients with hemophilic arthropathy.

Material and method. Multicenter cross-sectional cohort study. Eighty-eight patients will be recruited. The dependent variable will be physical activity (International Physical Activity Questionnaire). Secondary variables will be kinesiophobia (Tampa Kinesiophobia Scale), functionality (Functional Independence Scale in Hemophilia), pain intensity, and clinical, anthropometric, and sociodemographic variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemophilia A or B
* Over the age of majority
* With a medical diagnosis of severe phenotype of the disease
* With a medical diagnosis of hemophilic arthropathy in the lower limbs
* Under on-demand or prophylactic drug treatment.

Exclusion Criteria:

* Patients who require technical aids for walking
* Patients who are dependent for activities of daily living
* Patients over the age of 60
* Patients with cognitive impairments that prevent them from understanding the questionnaires

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with hemophilia A or B and hemophilic arthropathy where it is desired to assess the degree of physical activity and the main predictive factors for this.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2025-05-04 (Estimated); Primary Completion 2025-05-28 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
Measurement of physical activity level | Screening visit
  Physical activity levels will be assessed using the International Physical Activity Questionnaire (IPAQ). This tool assesses physical activity levels in adults aged 18 to 65. It consists of seven questions that ask about the frequency, duration, and intensity of physical activity performed in the last week. It also assesses the time spent walking and sitting. The results are classified into three categories: low, moderate, and high activity. The unit of measurement is metabolic equivalent task (METS), where a higher number of METS indicates greater physical activity.

SECONDARY OUTCOMES:
Measurement of fear of movement | Screening visit
  Fear of movement will be measured using the Tampa Kinesiophobia Scale (TSK). This self-reported questionnaire consists of 17 items, using a 4-point Likert scale. It comprises two subscales: avoidance of physical exertion due to fear of injury or pain, and belief that significant underlying medical problems exist. The total score ranges from 17 to 68 points, with a score of 37 or more indicating a high level of kinesiophobia
Measurement of degree of functional independence | Screening visit
  The degree of functional independence of patients will be measured using the Functional Independence Scale for Hemophilia (FISH). This tool measures eight activities of daily living: eating, personal hygiene, dressing, transferring from a chair, squatting, walking, climbing stairs, and running. Each activity is rated according to the level of assistance required, using a scale from 1 to 4. The total score can reach a maximum of 32 points, with a higher score indicating greater functional independence.
Measurement of the joint pain | Screening visit
  Pain intensity will be measured using the Visual Analog Scale (VAS). This is a simple and effective tool for measuring pain intensity. It consists of a horizontal line, usually 10 cm long, with one end representing "no pain" and the other "maximum pain imaginable."
Measurement of age | Screening visit
  The sociodemographic variable age will be measured in months completed from the date of birth
Measurement of marital status | Screening visit
  The sociodemographic variable marital status will be measured as a qualitative variable (single/married/divorced/widowed).
Measurement of educational level | Screening visit
  The sociodemographic variable educational level will be measured as a qualitative variable (primary education/secondary education/university education/vocational training).
Measurement of employment status | Screening visit
  The sociodemographic variable employment status will be measured as a qualitative variable (self-employed/employed by others/civil servant/unemployed/unable to work/retired).
Measurement of hemophilia type | Screening visit
  The clinical variable hemophilia type will be measured as a dichotomous variable (hemophilia A/hemophilia B).
Measurement of type of drug treatment | Screening visit
  The clinical variable drug treatment will be measured as a dichotomous variable (on-demand treatment/prophylactic treatment).
Measurement of inhibitor development | Screening visit
  The clinical variable development of antibodies prior to FVIII/FIX concentrates (inhibitors) will be measured as a dichotomous variable (yes/no).
Measurement of weight | Screening visit
  The anthropometric variable weight will be measured as a quantitative variable (measured in kg).
Measurement of height | Screening visit
  The anthropometric variable height will be measured as a quantitative variable (measured in cm).

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, Principal Investigator — Universidad de Oviedo
Locations (1):
- Universidad Católica San Antonio de Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No